CLINICAL TRIAL: NCT06612554
Title: Role of Zinc Supplementation in Immunological Non-responders HIV Individuals: Exploring Pathways for Persistent Inflammation
Brief Title: Zn Supplementation in HIV Immunological Non Responders
Acronym: VIHZn
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Hospital de Sabadell (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023/11335/I; PI23/00456 (Other Grant/Funding Number: ISCIII/FIS)
Record Dates: First submitted 2024-09-15; First posted 2024-09-25 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: HIV; Zinc Status; HIV Infection
Keywords: Zinc Supplementation; HIV Immunological Non-Responder; Immune response; immune activation; Inflammation
MeSH Terms: conditions — HIV Infections; Inflammation | interventions — Zinc Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablets will be administered. Three Tablets will be with the same shape and size that Zn supplement tablets during 16 weeks
  Interventions: Other: Placebo
- Zn Supplementation (Experimental): 16 weeks with 3 tablets of zinc (83mg Zinc acetate/tablet)
  Interventions: Dietary Supplement: zinc acetate

INTERVENTIONS:
Dietary Supplement: zinc acetate — Participants in Control group. They will continue the SoC + 3 tablets of placebo and participants in Zinc supplementation group. Tablets will be separated 12h (just in case the ART is based in Integrase Inhibitors (INSTI)) during supplementation for 16 weeks with 3 tablets of zinc (83mg Zinc acetate/tablet).
  Arms: Zn Supplementation
Other: Placebo — participants in Control group. They will continue the SoC + 3 tablets of placebo. 3 tablets separated 12h from ART during 16 weeks
  Arms: Placebo

SUMMARY:
Zinc is an essential micronutrient crucial for the normal functioning of the human immune system. Zinc deficiency impairs immune function and increases infection risk, especially in vulnerable populations like people living with HIV. This project aims to study the role of zinc supplementation in improving immune response in HIV-infected individuals who are Immunological Non-Responders (INRs)-people who have not restored Cluster of differentiation 4 (CD4) T-cell counts despite receiving antiretroviral therapy (ART). INRs face a higher risk of opportunistic infections, non-HIV comorbidities due to high inflammation, and generally have a poorer prognosis. Zinc supports immune function by aiding in immune cell development, cytokine production, and maintaining mucosal barrier integrity.

Several studies have investigated zinc supplementation in HIV-infected individuals, showing significant increases in CD4 counts and a reduction in opportunistic infections. However, the doses used vary, and the results are sometimes contradictory. Our objective is to study whether zinc supplementation in INRs improves immune function, specifically by increasing CD4 counts, decreasing inflammation, and affecting other immune parameters.

This project involves a clinical trial where INRs will be randomly assigned to receive 75mg of elemental zinc daily (in the form of 3 zinc acetate tablets) along with their usual treatment or to continue their treatment without zinc supplements. We will assess whether zinc supplementation increases CD4 lymphocytes, reduces inflammation in INRs, and induces immune system changes. We will also investigate immune system functionality by measuring the presence of the Torque Teno Virus (TTV), a harmless virus, and see how zinc supplementation impacts its control by monitoring viral load changes.

Recent research by our group has demonstrated that zinc has both antiviral and anti-inflammatory effects. Zinc supplementation is generally safe and well-tolerated, with few adverse effects. Zinc is available in various forms, including gluconate, acetate, and sulfate. Although the recommended daily dose is 40mg, studies have shown that doses exceeding 80mg have been safely administered for over 10 years without side effects.

We have selected a 75mg daily dose of elemental zinc for several reasons. Studies that showed no effect used lower doses (15-20mg/day), and our research found that 75mg/day improved outcomes in acute viral infections like Severe Acute Respiratory Syndrome-Coronavirus-2 (SARS-CoV2). We believe previous failures to show zinc's efficacy were due to insufficient dosing. After extensive literature review, we concluded that 75mg daily is safe and likely to produce the desired effects.

Our goal is to demonstrate the efficacy of zinc as an immunomodulatory agent. If successful, this could be a simple and cost-effective way to improve the quality of life for many people. We would recommend its widespread use under medical supervision, particularly at the doses being studied.

DETAILED DESCRIPTION:
Studies of people living with HIV show that although antiretroviral treatments (ART) decreases inflammation, a number of inflammatory markers remain persistently elevated and this chronic inflammation can play an important role in cardiovascular disease (CVD). Moreover, some individuals with HIV initiating ART do not recover Cluster of differentiation 4 (CD4+) T-cells count as expected, and are described as Immunological Non-Responders (INRs). INRs present with severely altered immunological functions, including malfunction and diminished production of cells within lymphopoietic tissue, perturbed frequencies of immune regulators such as regulatory T cells and Th17 cells, and increased immune activation, immunosenescence, and apoptosis. Importantly, INRs have an increased risk of morbidity and mortality compared to HIV-infected patients with an optimal immune reconstitution. Our group has demonstrated how this group responds poorly to messenger RNA (mRNA) vaccination against Severe Acute Respiratory Syndrome-Coronavirus-2 (SARS-CoV2) showing an impaired immune function among these individuals.

However, the definition of Immunological Non-Responders (INRs) suffers from lack of consensus impeding the comparison of findings. There seems to be agreement that an adequate immune response to antiretroviral treatment should include a CD4+ cells count more than 500 cells/μL, mainly because HIV-infected patients with this level of immune restoration have a morbidity and mortality rate approaching or comparable to those of HIV negative individuals. Patients with CD4+ cell counts <500 cells/μL are consequently classified as inadequate responders, included in the INRs group. And, although they are a group poorly described, their morbidity and mortality seem to be more similar to INRs than to adequate responders.

The underlying mechanism that explains INRs phenomena is not well understood. Several hypotheses have been raised as an older age, a long duration of HIV infection prior to antiretroviral treatment, co-infection with hepatitis C, and a low CD4 nadir predispose to immunological nonresponse. The CD4 nadir specifically appears to be critical for the recovery of CD4+ cells. However, none of these factors provide a full explanation for the lack of immune reconstitution in INRs. Probably this is the consequence of several factors and its interaction. Interestingly, low plasma zinc levels and inadequate zinc intake were found in up 50% of participants in several cohorts of HIV infected adults, and were independently associated with faster HIV disease progression and increased mortality. Zinc deficiency reduces generation of T-cells, depresses humoral and cell-mediated immunity, leads to lymphopenia, and thymic atrophy, and increases the frequency and number of infections. Thus, the zinc status could also have a role in the mechanisms involved in INRs.

Zinc in viral infection Zinc is an essential trace element for both host and pathogens. In order to grow, pathogens require zinc. Thus, zinc is a structural cofactor of viral proteins and certain viruses have developed strategies to alter cellular zinc homeostasis on its benefit. On the other hand, there is extensive evidence that zinc can prevent viral replication and lower cellular invasion (eg. Rhinovirus, Hepatitis C,SARS-CoV2).

Remarkably, our team has shown that low zinc levels favor SARS-CoV2 expansion. These results might indicate either a direct anti-viral action against SARS-CoV2 or that the virus benefits from stress conditions caused by low levels of cellular zinc. Zinc supplementation has been shown to be beneficial when administering to Hepatitis B and Hepatitis C infected patients. Moreover, zinc-based nutritional immunity reduces diarrheal episodes and respiratory tract diseases. Remarkably, zinc supplementation for the common cold caused by rhino- and coronaviruses prevents it and reduces its duration, if the administration starts within 24h after the onset of symptoms. Thus, zinc supplementation has been proven beneficial against some viral infections. However, whether this was caused by improved local immune response or viral inhibition remains uncertain.

Zinc as immunomodulator Zinc deficiency (ZD) is known to be associated with proinflammatory responses at infection, showing higher reactive oxygen species (ROS) production and inflammatory markers. An imbalance in cytokine production by cells of both innate and adaptive immunity has also been reported.

Concretely, ZD is associated with higher levels of Interleukin-6 (IL-6), Interleukin-1beta (IL-1beta) and Tumor Necrosis Factor-alpha (TNF-a). In this scenario, zinc supplementation has been shown to decrease the incidence of infection, inflammatory cytokines, including IL-6, and oxidative stress markers in elderly individuals. Moreover, zinc supplementation has been shown to balance immune responses.

Nutritional zinc status and IL-6 are highly interconnected. Thus, IL-6 can reduce zinc bioavailability promoting internalization in hepatocytes and the expression of zinc chelators. On the other hand, zinc decreases IL-6 production via inhibition of Signal Transducer and Activator of Transcription-3 (STAT-3) pathway. Our study with Coronavirus Disease-19 (COVID-19) patients showed a negative correlation between serum zinc levels and IL-6 production.

Zinc in T lymphocytes activation and exhaustion Zinc is known to affect T lymphocyte maturation, differentiation and cytokine production. Activated T cells are known to increase zinc content. On the one hand, zinc has been shown to be required for the correct T-cell Receptor (TCR) signaling by modulating Lck and Zap- 70 activity. Our collaborators Vicente et al. have demonstrated that zinc positively potentiates the three main signaling pathways, Nuclear Factor-kB (NF-kb) and Nuclear Factor of Activated T-cells-1. The knock-down of Zip6, a zinc transporter up regulated early during cell activation, alters zinc entry and dramatically impairs activation of Jurkat T cells. Moreover, recent studies on Cluster of differentiation 8 (CD8) T-cell dysfunction during cancer and chronic infections have started to elucidate the transcriptional pathways involved in this phenomenon and zinc homeostasis has emerged again as a key element. Thus, metallothioneins 1 and 2 levels and zinc dependent transcription factors are differentially expressed in exhausted CD8+ cells. Nonetheless, there are no studies investigating whether zinc supplementation/chelation might directly affect the CD8+ dysfunctional profile and how these learnings could be translated into novel therapeutic approaches for these diseases including HIV infection.

Zinc in B lymphocyte function It has been shown that zinc transporters (Zip7 and Zip10) are essential in B cell function. B cells activation and plasma cell differentiation depends on zinc signaling. Nutritional zinc status is an important factor determining antibody production given its action on both, B-cells and CD4+ T lymphocytes. Thus, ZD has been shown in mouse models to lower humoral immune response.

Preliminary Results Our group has been working in the immunomodulatory effect of zinc in viral infections and in the immune response since 2020. Also, we are actively working in the immune response in people with HIV (PWH) INRs. We have several publications and an active research line putting these two research lines together.

We previously carried out a study analyzing the association between zinc plasma levels at hospital admission and COVID-19 prognosis, during the first wave of the pandemics. We found a negative correlation between the zinc levels and IL-6, as well as with mortality. We also found that zinc acted on viral replication in vero cell cultures. We have recently conducted a clinical trial (NCT05778383) whose preliminary results have been reported in CROI2023 #542. In this trial, we observed that high-dose Zinc supplementation in the acute phase of SARS-coV-2 infection is associated with a better prognosis of the disease. We also shown an abnormal immune response to vaccination among INRs. Therefore, we have demonstrated in a viral infection context that zinc has an antiviral and anti-inflammatory effect, which may have a benefit in people living with HIV, especially in the INR situation.

Hypothesis

This study has several hypotheses:

1. Relative low zinc levels are frequent in our cohort of HIV patients and have a role in worse immune response and in higher inflammatory response.
2. We hypothesize that zinc has an impact in the immune system restoring the lymphocyte count in INRs HIV individuals and improving immune function and inflammation associated with chronic viral infection.

   Therefore, zinc supplementation in physiological concentrations and recommendations has a beneficial impact in immune function, reducing immune activation and reducing chronic inflammation in INRs HIV individuals.
3. Zinc supplementation protects gut mucosa of cytopathic effect of virus, restoring partially the gut permeability induced by HIV
4. Zinc supplementation improves oxidative stress and mitochondrial function

Objectives

The main objective is to study the clinical and immune benefits of 16 weeks of supplementation with zinc acetate in HIV immunological non-responders individuals. To address this objective, a Randomized Clinical Trial (RCT) will be designed.

Aim 1: To design an double blinded randomized multicentric 2-arm study The following parameters will be measured at baseline and at week-16 in zinc-supplemented individuals vs controls:

* Primary: Change in CD4+ T-cell count
* Secondary: Changes in Quality of life changes through EuroQol-5D-3L, CD4+ CD8+ T-cell activation, T-cell subsets, Torque Teno Virus replication, IL-6, C-RP, Transcriptomics, ROS

Aim 2. To measure persistence in changes quality of life, immune function, immune activation, inflammatory biomarkers, and mitochondrial function and ROS at week 24 respect to week-16 and baseline. In terms of: Changes in Quality of life changes through EuroQol-5D-3L, CD4+ CD8+ T-cell activation, T-cell subsets, Torque Teno Virus replication, IL-6, C-RP, Transcriptomics, ROS

The methodology is divided into tasks.

Task 1. Randomized Clinical Trial. An open label randomized multicentric 2-arm study will be designed. Participants will be prospectively enrolled at two sites Hospital del Mar and Hospital Parc Taulí. In the Zinc Supplementation group (Zn), participants will received the Standard of Care (SoC) and separated 12h (just in case the ART is based in Integrase Inhibitors (INSTI)) will be supplemented during 16 weeks with 75mg of elemental Zn (3 tablets (83mg Zn acetate) 249mg of Zinc Acetate Zinc-NM; Laboratorios Cantabria (Spanish National Code 156252.4)). We have selected 75mg of elemental Zn/d as oral supplementation because it has been used safely in non-HIV studies with 1 year duration at this concentration with no serious adverse effects (15). End of Treatment (EoT) will be at 16 weeks, but a follow up up to 24-weeks will be done to assess the persistence of the effects of Zn.

The study involves multiple tasks across different visits and sample collections, aiming to assess the effects of the intervention on immune response, inflammation, and oxidative stress in participants.

Task 1.1: Visits and Sample Collection

Participants will undergo three visits:

Visit 1 (Screening/Randomization/Baseline): In-person visit where randomization is performed using REDCap. After informed consent, medical history is recorded, vital signs are taken, and blood samples are collected for various tests, including CD4+ T-cell count, HIV viral load, C-reactive protein (CRP), ferritin, D-dimer, vitamin D, and zinc. Participants also complete the EuroQol-5D-3L quality of life questionnaire. Blood samples are collected in serum, ethylenediaminetetraacetic acid (EDTA), and RNA tubes for peripheral blood mononuclear cells (PBMCs).

Visit 2 (Week 16): Similar assessments as Visit 1 are performed, with the addition of tracking adverse events (AEs) and concomitant therapies.

Visit 3 (Week 24): The same tests are repeated to extend the study, with sample collection focusing on the same biomarkers as in prior visits.

Task 2: T-cell Subset Assessment PBMCs from the enrolled participants will be isolated using density gradient centrifugation. Samples are preserved at -80°C and sent to IMIM for processing. Flow cytometry will be used to analyze T-cell subsets, including markers like CD45, CD4, CD8, FOXP3, and PD-1, with data analyzed using FlowJo software.

Task 3: Multiplex ELISA for Inflammatory Biomarkers At baseline, Week 16, and Week 24, fasting blood sera will be collected to measure inflammatory markers such as sCD14, sCD163, CRP, sTNFR-I, sTNFR-II, and gut integrity markers like IFABP and Lipopolysaccharide-binding protein (LBP), using ELISA.

Task 4: Torque Teno Virus (TTV) Viral Load TTV viral load will be quantified using the TTV R-GENE kit, with DNA extracted and analyzed via TaqMan real-time Polymerase Chain Reaction (rt-PCR) at baseline, Week 16, and Week 24.

Task 5: ROS and Mitochondrial Function Reactive Oxygen Species (ROS) are chemically reactive molecules containing oxygen, such as free radicals and peroxides. They are byproducts of cellular metabolism and play essential roles in cell signaling and homeostasis. However, excessive ROS can cause oxidative stress, damaging DNA, proteins, and lipids, which can lead to various diseases, including cardiovascular diseases, neurodegeneration, and cancer.

To assess ROS levels, indirect markers such as glutathione (GSH/GSSG ratio), 4-hydroxynonenal (4-HNE), and malondialdehyde (MDA) are commonly measured. Glutathione helps neutralize ROS, with its GSH/GSSG ratio indicating oxidative stress. 4-HNE and MDA are byproducts of lipid peroxidation, providing insights into cellular membrane damage due to ROS. These markers are typically measured using techniques like enzymatic assays, ELISA, and TBARS assay, respectively. Understanding ROS levels and their effects is critical for studying oxidative stress and related diseases.

Task 6: Transcriptomic Analysis RNA will be extracted from blood samples at baseline and Week 16 for transcriptomic analysis using expression microarrays. Bioinformatics analysis will be conducted at the MARGenomics platform to study gene expression changes related to the intervention.

B.-Secondary outcomes

1.-Change in the transcriptome profile between baseline and week 16 respect to week 24 in whole blood samples

C.-Safety endpoints

-Incidence of adverse events (AEs)

ELIGIBILITY:
Inclusion Criteria:

* confirmed HIV infection;
* 18 years or older
* Serum zinc levels less than 150ug/dl (normal range considered 75-150 ug/dl)
* HIV-1 infection on stable ART for at least 3 months with cumulative ART duration of at least 6 months
* Undetectable (less than 50copies/ml) persistently (isolated transient increases in viremia of less than 1000 copies/ml will be accepted)
* Persistent less than 500CD4+ T-cells/mm3 at enrolment or an increase of less than 80 cells/mm3 after one year of viral undetectability

Exclusion Criteria:

* Pregnancy
* Lactation
* Active infectious or inflammatory condition
* Uncontrolled diabetes
* Serum Zinc levels more than 150ug/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
CD4+ T-cell number change | 16 weeks
  CD4+ T-cell count (cells/ml)

SECONDARY OUTCOMES:
Change in CD4+Tcell activation | 16 weeks
  change in % CD38+ CD4+ T-cell
Change in CD8+Tcell activation | 16 weeks
  change in % CD38+ CD8+ T-cell
Change in Quality of Life EuroQol-5D-3L | 16 weeks
  Quality of life changes through EuroQuality of life-5D-3L (EuroQol-5D-3D). Highest (best Quality of life) 1.minimum value (less or equal to 0-worse quality of life)
Changes in Interleukin-6 | 16 weeks
  Changes in Interleukin-6 (pg/mL)
Changes in C-Reactive protein | 16 weeks
  Changes in C-Reactive-Protein (mg/dl)
Changes in ROS by malondialdehyde | 16 weeks
  Measure changes in malondialdehyde in nmol/mL through Lipid Hydroperoxide Assay
Changes in ROS induced lipid peroxidation by 4-hydroxynonenal | 16 weeks
  Measure changes 4-hydroxynonenal by ELISA (nmol/mg protein)
Changes in ROS by gluthathione production | 16 weeks
  Measure changes in glutathione by gluthathione Assay (GSH/GSSG) (nmol/mg protein)
Transcriptomic changes | 16 weeks
  Analyze gene expression changes in inflammatory pathways through RNA sequencing and qPCR to assess oxidative stress-induced inflammation
Torque Teno Virus viral load | 16 weeks
  Measure Torque Teno Virus by quantitative Polymerase Chain Reaction (qPCR)

OTHER OUTCOMES:
Changes at week 24 CD4+ T-cell number change | Week 24
  Changes in total CD4+ T-cell count (cells/ml) 8 weeks after stopping supplementation.
Changes at week 24 CD4+Tcell activation | Week 24
  change in % CD38+ CD4+ T-cell at week 24
Changes at week 24 CD8+Tcell activation | Week 24
  change in % CD38+ CD8+ T-cell at week 24
Changes at week 24 in Quality of Life EuroQol-5D-3L | Week 24
  Quality of life changes through EuroQuality of life-5D-3L (EuroQol-5D-3D). Highest (best Quality of life) 1.minimum value (less or equal to 0-worse quality of life)
Changes in Transcriptomic at week 24 | Week 24
  Analyze gene expression changes in inflammatory pathways through RNA sequencing and qPCR to assess oxidative stress-induced inflammation
Changes in ROS by malondialdehyde at week 24 | Week 24
  Measure changes in malondialdehyde in nmol/mL through Lipid Hydroperoxide Assay
Changes in ROS by changes in 4-hydroxynonenal at week 24 | Week 24
  Measure changes 4-hydroxynonenal by ELISA (nmol/mg protein)
Changes in ROS by changes in gluthathione at week 24 | Week 24
  Measure changes in glutathione by Glutathione Assay (GSH/GSSG) (nmol/mg protein)

IPD SHARING:
Plan to Share IPD: Undecided
We will provide the IPD upon reasonable request to the PI

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/54/NCT06612554/SAP_000.pdf